CLINICAL TRIAL: NCT06481943
Title: A Prospective Research Investigation of Ischemia Using SandboxAQ Magnetocardiography Device
Brief Title: A Prospective Research Investigation of Ischemia Using MCG
Acronym: PRISM/PRISM2
Status: Recruiting | Type: Observational
Sponsor: SB Technology, Inc. (Industry)
Collaborators: Mayo Clinic (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: SB-ACS-003, SB-ACS-005
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Acute Coronary Syndrome
Keywords: Magnetocardiography; MCG
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- ACS: Adult patients who are undergoing a diagnostic angiography or revascularization procedure for the diagnosis or treatment of ischemia or acute coronary syndrome (ACS). Patients are further classified as having low, medium, and high risk for ACS.
  Interventions: Device: Sponsor MCG device (CardiAQ)

INTERVENTIONS:
Device: Sponsor MCG device (CardiAQ) — Unshielded magnetocardiography device for measuring cardiac magnetic fields

SUMMARY:
PRISM is a prospective, pilot research study that aims to systematically characterize the usefulness of CardiAQ MCG, a bedside magnetocardiography device, in the evaluation of myocardial ischemia and infarction status.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo a diagnostic angiography or revascularization procedure for the diagnosis or treatment of ischemia or acute myocardial infarction
* Ability for participant to comply with study requirements
* Patient consented before the planned, clinically indicated cath-lab procedure begins to allow sufficient time for study related activities
* Written informed consent

Exclusion Criteria:

* Present STEMI
* Pregnant or breastfeeding
* Having an active atrial fibrillation episode as seen on most current 12-lead ECG
* Active thoracic metal implant
* Poor access to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are undergoing a diagnostic angiography or revascularization procedure for the diagnosis or treatment of ischemia or acute coronary syndrome (ACS).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Relationship between pre-procedural MCG and the peri-procedural angiography-based measures | Data taken within 24 hours of each other
  Utilize linear regression and logistic regression to determine whether a set of a priori MCG-based biomarkers can prospectively predict the objective clinical assessment of ACS, while statistically adjusting for covariates.

SECONDARY OUTCOMES:
Sponsor MCG device safety | 30 days
  Device-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kit Yee Au-Yeung, PhD, Study Director — SB Technology, Inc.
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai Hospital, New York, New York